CLINICAL TRIAL: NCT07071792
Title: Prevalence of Helmet Associated Neck Pain Among Tcs Riders
Status: Completed | Type: Observational
Sponsor: Elite College of Management Sciences, Gujranwala, Pakistan (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-GCUF-079260
Record Dates: First submitted 2025-07-06; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Neck Pain
Keywords: Helmet use; neck pain; motorcycles; head protective devices; disability
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim and objective of this study is to check the prevalence of helmet associated neck pain among TCS riders.

DETAILED DESCRIPTION:
Finding the overall prevalence of neck pain linked to helmet use is the goal of the study. On the other hand, the TCS delivery riders of Gujranwala, who wear helmets for extended periods of time throughout their daily employment, are a larger and more pertinent demographic in our study. Furthermore, our study is a significant and much-needed addition to this field as no prior research has explicitly examined the prevalence of helmet-associated neck pain among TCS riders.

ELIGIBILITY:
Inclusion Criteria:

* 18-45-year age
* male TCS riders
* All TCS riders who are using helmet for past six months or above
* Minimum duration of helmet use
* who will be willing to participate

Exclusion Criteria:

* Subjects had any known disorder that causes pain in neck or upper limb
* Any traumatic injury to cervical spine (fractures)
* cervical spine pathologies

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Males were selected for this study because, in Pakistan, the occupation of TCS rider is predominantly held by men. Therefore, to ensure relevance and accuracy, the study population was limited to male participants
Study Population: TCS riders who use helmets for at least 6 hours per day
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 12 weeks
  to measure helmet associated neck disability, ranging from 0 (no disability) to 50 (complete disability)
Numeric Pain Rating Scale | 12 weeks
  to measure helmet associated neck pain, high score indicates worse patient condition

CONTACTS AND LOCATIONS:
Overall Officials: Syeda Mahnoor Hassan, MSPT, Principal Investigator — Elite College of ManagementSciences
Locations (1):
- TCS centers, Gujranwala, Punjab Province, Pakistan

REFERENCES:
- [Background] Makkiyah FA, Natashia K, Kristanti M, Purwaningastuti DA. Associated Factors with Neck Pain among Productive Adult Motorcyclists in Metropolitan University Settings : A Cross-Sectional Study. J Korean Neurosurg Soc. 2025 Jul;68(4):425-435. doi: 10.3340/jkns.2024.0114. Epub 2024 Nov 26. PMID 39591956
- [Background] Harrison MF, Forde KA, Albert WJ, Croll JC, Neary JP. Posture and Helmet Load Influences on Neck Muscle Activation. Aerosp Med Hum Perform. 2016 Jan;87(1):48-53. doi: 10.3357/AMHP.4301.2016. PMID 26735233